CLINICAL TRIAL: NCT03168737
Title: Test-Retest of (18)F-Fluoroazomycin Arabinoside ([18F]FAZA) PET-CT of Solid Tumors
Brief Title: 18F-Fluoroazomycin Arabinoside PET-CT in Diagnosing Solid Tumors in Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0847; NCI-2018-01196 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0847 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Malignant Breast Neoplasm; Malignant Colorectal Neoplasm; Malignant Pancreatic Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms | interventions — fluoroazomycin arabinoside; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (18F-fluoroazomycin arabinoside, PET-CT scans) (Experimental): Patients receive 18F-fluoroazomycin arabinoside IV and after 60 minutes undergo 5 PET-CT scans at 60, 90, 120, 150, and 180 minutes on days 1 and 2.
  Interventions: Procedure: Computed Tomography; Radiation: Fluorine F 18-fluoroazomycin Arabinoside; Procedure: Positron Emission Tomography
- Group B (18F-fluoroazomycin arabinoside, PET-CT scans) (Experimental): Patients receive 18F-fluoroazomycin arabinoside IV and after 60 minutes undergo 5 or less PET-CT scans on day 1 and 5 or less PET-CT scans >= 24 hours later up to 10 days.
  Interventions: Procedure: Computed Tomography; Radiation: Fluorine F 18-fluoroazomycin Arabinoside; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET-CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Radiation: Fluorine F 18-fluoroazomycin Arabinoside — Given IV
  Other Names: 18F-FAZA; 18F-Fluoroazomycin Arabinoside; FAZA F-18; FLUOROAZOMYCIN ARABINOSIDE F-18
Procedure: Positron Emission Tomography — Undergo PET-CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This early phase I trial studies how well 18F-fluoroazomycin arabinoside positron emission tomography (PET)-computed tomography (CT) works in diagnosing solid tumors. Using 18F-fluoroazomycin arabinoside with PET-CT may help doctors plan better treatment for patients with solid tumors. 18F-fluoroazomycin arabinoside may help to show how much oxygen is present in a tumor during a PET-CT scan.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of PET-CT using 18F-fluoroazomycin arabinoside ([18F]FAZA) and to determine the optimal imaging time to detect hypoxia in solid tumors.

SECONDARY OBJECTIVES:

I. To determine the variability of imaging findings from repeated [18F]FAZA PET-CT studies over >= 24 hours up to 10 days.

II. To confirm the safety of [18F]FAZA administered during PET-CT imaging of hypoxia of solid tumors.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP A: Patients receive 18F-fluoroazomycin arabinoside intravenously (IV) and after 60 minutes undergo 5 PET-CT scans at 60, 90, 120, 150, and 180 minutes on days 1 and 2.

GROUP B: Patients receive 18F-fluoroazomycin arabinoside IV and after 60 minutes undergo 5 or less PET-CT scans on day 1 and 5 or less PET-CT scans >= 24 hours later up to 10 days.

After completion of study treatment, patients are followed up at 24 hours and at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologic diagnosis of a solid tumor. All solid tumors will be considered, but patients with breast, pancreas, and colorectal masses will be prioritized.
* Patient must have a solid tumor with a short-axis greater than or equal to 1 cm (by CT, magnetic resonance imaging [MRI], ultrasonography or mammography) to allow reliable PET imaging.
* A patient who has not received systemic or loco-regional treatment of the tumor within the last month.
* Ability of the subject, or the legally authorized representative (LAR) if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable, to understand, and the willingness to sign, a written informed consent.
* Patients who are not expected to receive cancer therapy before imaging sessions are completed.

Exclusion Criteria:

* Pregnant or lactating women: pregnant women are excluded from this study because the effects of [18F] FAZA in pregnancy are not known. A urine or serum pregnancy test will be performed before accrual after informed consent is obtained.
* Lactation should be suspended for at least two days following the administration of [18F] FAZA to the mother, because of the unknown but potential risk for adverse events in nursing infants secondary to administration of the radionuclide to a lactating woman.
* Subjects with contraindications to the use of [18F] FAZA including confirmed allergy.
* Patients with a body weight of 400 pounds or more, or a body mass index (BMI) which precludes their entry into the bore of the PET/CT scanner, because the findings will probably be compromised in image quality with CT, PET/CT and MRI.
* Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the investigator may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Relative change of imaging parameters (tumor volume, standardized uptake value [SUV], tumor to muscle ratio [TMR], hypoxic tumor volume [HTV1, HTV2], and total lesion hypoxia [TLH1, TLH2]) | Baseline up to 30 days
  Summary statistics of tumor volume, SUV, TMR, HTV1, HTV2, TLH1, TLH2, and their changes from baseline to later time point will be provided in mean, standard deviation, and range by time point. Lin's concordance correlation coefficient for these parameters will be calculated and MDC95 will also be calculated for 2 hour timepoint or other time points. Other statistical analyses will be carried out as appropriate.
Incidence of adverse events per Common Terminology Criteria for Adverse Events version 4.03 | Up to 30 days
  Adverse events and vital signs will be monitored and described with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Franklin C Wong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org